CLINICAL TRIAL: NCT05741788
Title: The Teaspoon Study - Telefitting Spinal Cord Stimulation for Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Teaspoon
Record Dates: First submitted 2023-01-16; First posted 2023-02-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Chronic Pain
MeSH Terms: conditions — Spinal Cord Injuries; Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Prospective cohort of patients clinically scheduled to undergo spinal cord stimulation for the treatment of chronic back pain or radiculopathy.
  Interventions: Device: Various Stimulation Patterns

INTERVENTIONS:
Device: Various Stimulation Patterns — Participants will undergo a structured optimization evaluating existing types of stimulation (tonic, burst, and multistim). Each participant will try out all types of available stimulation but be blinded to the type. Over the course of four months, each participant will evaluate each type of stimulation by reporting daily pain scores. Participants will follow up routinely to collect laboratory, behavioral, and survey responses to test for the feasibility of obtaining data explaining pain phenotype.

SUMMARY:
Spinal cord stimulation modulates the nervous system to effectively block pain signals originating from the back and legs. Spinal cord stimulation has been shown to improve chronic pain, improve quality of life, and reduce disability. Unfortunately, spinal cord stimulation has a high trial failure rate and a high long-term failure rate. This study consists of a prospective cohort of patients clinically scheduled to undergo spinal cord stimulation for the treatment of chronic back pain or radiculopathy. Participants will undergo a structured optimization evaluating existing types of stimulation (tonic, burst, and multistim). Each participant will try out all types of available stimulation but be blinded to the type. Over the course of four months, each participant will evaluate each type of stimulation by reporting daily pain scores. Thompson sampling will be used to identify which setting produces the biggest improvement in pain and recommend it for future use. Participants will follow up routinely to collect laboratory, behavioral, and survey responses to test for the feasibility of obtaining data explaining pain phenotype.

ELIGIBILITY:
Inclusion Criteria:

* 22 years of age or older
* Scheduled to undergo spinal cord stimulation
* English speaker
* Baseline pain rating (NRS/VAS) >=6

Exclusion Criteria:

* Scheduled for permanent implantation only without trial
* Presence of pacemakers or other neurostimulators
* Pregnant
* Inability to read or use smart phone
* Individuals who are unable to consent
* Employees or students of PI
* Prisoners

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility | 3 years
  Feasibility as measured by total study procedure completion rate.

SECONDARY OUTCOMES:
Acceptability of procedure | 3 years
  Acceptability as measured by the average patient rating and their acceptability of the study based on their experience during the procedures across study procedures. Participants rate their overall experience with the procedures used during the study on a scale from 0 as 'Excellent' to 4 as 'Very Poor'.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No